CLINICAL TRIAL: NCT00536991
Title: A Phase I/II Study of Oral Calcitriol in Combination With Ketoconazole in Androgen Independent Prostate Cancer
Brief Title: Calcitriol in Combination With Ketoconazole and Therapeutic Hydrocortisone in Treating Patients With Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: difficult to recruit
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 68905; NCI-2011-00129 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RPCI-I-68905; I 68905 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Prostate Adenocarcinoma; Recurrent Prostate Carcinoma; Stage III Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Calcitriol; Ketoconazole; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (calcitriol, ketoconazole, hydrocortisone) (Experimental): PHASE I: Patients receive calcitriol PO QD on days 1-3, 8-10, 15-17, and 22-24. Patients also receive ketoconazole PO TID on days 1-24 and therapeutic hydrocortisone PO BID on days -1 to 24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients receive calcitriol and therapeutic hydrocortisone as in phase I. Patients also receive ketoconazole PO TID on days 4-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: Calcitriol; Drug: Ketoconazole; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Therapeutic Hydrocortisone

INTERVENTIONS:
Dietary Supplement: Calcitriol — Given PO
  Other Names: 1,25(OH)2-D3; 1,25-Dihydroxycholecalciferol; Calcijex; Rocaltrol
Drug: Ketoconazole — Given PO
  Other Names: Fungarest; Fungoral; Ketoderm; Ketoisdin; Nizoral; Orifungal M; Panfungol; R-41400; Xolegel
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Therapeutic Hydrocortisone — Given PO
  Other Names: Aeroseb-HC; Barseb HC; Barseb-HC; Cetacort; Cort-Dome; Cortef; Cortenema; Cortifan; Cortisol; Cortispray; Cortril; Dermacort; Domolene; Eldecort; Hautosone; Heb-Cort; HYDROCORTISONE; Hydrocortone; Hytone; Komed-HC; Nutracort; Proctocort; Rectoid

SUMMARY:
This phase I/II trial studies the side effects and best dose of calcitriol when given in combination with ketoconazole and therapeutic hydrocortisone and to see how well it works in treating patients with prostate cancer. Calcitriol may help prostate cancer cells become more like normal cells and grow and spread more slowly. Ketoconazole and therapeutic hydrocortisone may help calcitriol work better by making tumor cells more sensitive to the drug. Giving calcitriol together with ketoconazole and therapeutic hydrocortisone may be a better treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of oral calcitriol daily x 3 consecutive days a week in combination with oral ketoconazole (400 mg thrice daily [TID]) + oral hydrocortisone (20 mg AM, 10 mg PM) in men with androgen independent prostate cancer (AIPC). (Phase I) II. To estimate the prostate-specific antigen (PSA) response rate. (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of the phase II dose of oral calcitriol with and without ketoconazole (400 mg TID).

II. Describe any objective tumor responses to the combination of oral calcitriol and ketoconazole and hydrocortisone among patients with measurable disease using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

III. Determine toxicities and tolerability of oral calcitriol combination with daily oral ketoconazole and hydrocortisone.

OUTLINE: This is a phase I, dose-escalation study of calcitriol followed by a phase II study.

PHASE I: Patients receive calcitriol orally (PO) once daily (QD) on days 1-3, 8-10, 15-17, and 22-24. Patients also receive ketoconazole PO TID on days 1-24 and therapeutic hydrocortisone PO twice daily (BID) on days -1 to 24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients receive calcitriol and therapeutic hydrocortisone as in phase I. Patients also receive ketoconazole PO TID on days 4-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma consistent clinically with androgen independent prostate cancer
* Measurable disease with elevated PSA or evaluable disease (PSA elevation will constitute evaluable disease)
* =< 2 regimens of cytotoxic chemotherapy prior to study entry; retinoids, vitamin D analogues, peroxisome proliferator-activated receptor (PPAR) gamma agonists or antagonists, antiandrogens, progestational agents, estrogens, prostate cancer (PC)-SPES, luteinizing hormone-releasing hormone (LHRH)-analogues, vaccines, cytokines will not be considered "cytotoxics"; patients who have previously received ketoconazole + glucocorticoids will be eligible for this trial
* Patients who have received antiandrogens or progestational agents as therapy for prostate cancer must discontinue therapy and demonstrate a rising PSA >= 28 days following discontinuation (antiandrogen withdrawal- AAW) (>= 42 days for bicalutamide or nilutamide); patients who receive megestrol acetate as therapy for "hot flashes" at a dose of =< 40 mg per day may continue this therapy during this trial; the dose of the megestrol acetate should not be changed during protocol treatment; patients undergoing androgen deprivation using LHRH analogues must continue such agents or undergo orchiectomy to maintain castrate levels of testosterone
* Patients must have prostate cancer that is advanced or recurrent and for which standard curative or reliable palliative therapies do not exist or are no longer effective
* Patients should not have received any chemotherapy or investigational agents for at least 4 weeks before entering the study (6 weeks for nitrosoureas or mitomycin C)
* Eastern Clinical Oncology Group performance status =< 2 (Karnofsky >= 60%)
* Life expectancy > 3 months
* Leukocytes: >= 3,000/ul
* Hemoglobin: >= 8 g/dl
* Absolute neutrophil count (ANC): >= 1,500/ul
* Platelets: >= 75,000/ul
* Total bilirubin: within normal institutional limit
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT): =< 2.5 x institutional upper limit of normal
* Creatine: =< 2 mg/dL
* Calcium: not above normal institutional limit
* Patients should be able to receive oral medications
* Patients with brain metastases which are stable and have been treated with surgery or irradiation will be eligible for this trial
* Men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while her partner is participating in this study, she should inform the treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* PHASE II - GROUP B: Progressive disease must have occurred on abiraterone within the prior 12 months and patient has not received treatment with enzalutamide
* Men of all ethnic groups are eligible for this trial; efforts will be made to include minority groups and all representative ethnicities and races in the community serviced by Roswell Park Cancer Institute (RPCI)

Exclusion Criteria:

* Known severe hypersensitivity to ketoconazole, calcitriol or any of the excipients of these products
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to calcitriol, ketoconazole, or other agents used in study
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the trial
* History of kidney, ureteral, or bladder stones within the last 5 years
* Heart failure or significant heart disease including significant arrhythmias, myocardial infarction within the last 3 months, unstable angina, documented ejection fraction < 30%, or current digoxin therapy
* Thiazide therapy within 7 days from entering the study
* Requirement for concurrent systemic glucocorticoid therapy at greater than physiologic replacement doses
* Unwillingness to stop calcium supplementation
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease) or intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would lit compliance with study requirements
* Human immunodeficiency virus-positive patients receiving combination anti-retroviral therapy are excluded from the study
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, or St John's wort, alfentanil, alfuzosin, almotriptan, alprazolam, amiodarone, amitriptyline, amprenavir, aprepitant, aripiprazole, bepridil, bortezomib, bosentan, budesonide, buprenorphine, buspirone, carbamazepine, cilostazol, cisapride, cyclosporine, delavirdine, didanosine, digoxin, disopyramide dofetilide, donepezil, eletriptan, eplerenone, fluticasone, fosamprenavir, galantamine, systemic griseofulvin, indinavir, levobupivacaine, lopinavir, midazolam, mifepristone, modafinil, nateglinide, nefazodone, nelfinavir, oxcarbazepine, pimozide, quetiapine, quinidine, repaglinide, rifabutin, rifampin, rifapentine, ritonavir, saquinavir, sildenafil, sirolimus, tacrolimus, tadalafil, tolterodine, theophyllines, tolterodine, triazolam, valdecoxib, vardenafil, ziprasidone, zonisamide, statins, with the exception of pravastatin (Pravachol) or other "statins" which are not metabolized by or induce cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4), calcium channel blockers, Coumadin and macrolides or other agents that will be significantly perturbed in a clinically important way by the P450 inhibitory properties of ketoconazole
* Concomitant use of proton pump inhibitors or histamine (H)2 blockers
* Treatment with a non-approved or investigational drug or agent within 30 days before day 1 of trial treatment
* Any unresolved chronic toxicity greater then Common Terminology Criteria (CTC) grade 2 from previous anticancer therapy
* Incomplete healing from previous oncologic treatments or other major surgery
* Inability to swallow oral capsules
* Patients on digoxin will be excluded from this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saby George, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I/II: Oral Calcitriol, Ketoconazole, Hydrocortisone: oral calcitriol daily x 3 consecutive days a week in combination with oral ketoconazole, (400 mg TID) + oral hydrocortisone (20mg AM, 10mg PM) in men with androgen independent prostate cancer (AIPC).
Period: Overall Study
Arm/Group | Phase I/II: Oral Calcitriol, Ketoconazole, Hydrocortisone
Started | 51
Completed | 38
Not Completed | 13
Not completed — Withdrawal by Subject | 10
Not completed — Physician Decision | 1
Not completed — patient ineligible | 2

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Phase I/II: Oral Calcitriol, Ketoconazole, Hydrocortisone
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 45
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Determine the Maximum Tolerated Dose (MTD)
Description: Determine the maximum tolerated dose (MTD) of oral calcitriol daily x 3 consecutive days a week in combination with oral ketoconazole (400 mg thrice daily [TID]) + oral hydrocortisone (20 mg AM, 10 mg PM)
Time Frame: up to 11 years
Population: All Phase I participants
Measure: Number; unit: mcg
Groups:
- Treatment (Calcitriol, Ketoconazole, Hydrocortisone): PHASE I: Patients receive calcitriol PO QD on days 1-3, 8-10, 15-17, and 22-24. Patients also receive ketoconazole PO TID on days 1-24 and therapeutic hydrocortisone PO BID on days -1 to 24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  PHASE II: Patients receive calcitriol and therapeutic hydrocortisone as in phase I. Patients also receive ketoconazole PO TID on days 4-24. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Calcitriol: Given PO
  Ketoconazole: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Therapeutic Hydrocortisone: Given PO
Arm/Group | Treatment (Calcitriol, Ketoconazole, Hydrocortisone)
Number analyzed (Participants) | 14
mcg | 10

2. Primary Outcome: PSA Response Rate
Description: Patients will be considered evaluable for PSA response if they have at least two post-baseline PSA measurements at least 4 weeks apart, or if they have other evidence of disease progression. A PSA response will be considered a PSA decline of at least 50% must be confirmed by a second PSA value four or more weeks later. The reference PSA for these declines should be a PSA measured within 2 weeks prior to the initiation of therapy.
Time Frame: Up to 11 years
Population: All treated and eligible patients
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I/II: Oral Calcitriol, Ketoconazole, Hydrocortisone
Number analyzed (Participants) | 51
percentage of participants | 35 [22 to 50]

3. Secondary Outcome: Incidence of Toxicity Graded According to the National Cancer Institute CTC Version 3.0
Description: Count of participants with serious adverse event. Please refer to the adverse event reporting for more detail.
Time Frame: Up to 11 years
Population: All treated and eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I/II: Oral Calcitriol, Ketoconazole, Hydrocortisone
Number analyzed (Participants) | 51
Participants | 14

4. Secondary Outcome: Objective Tumor Response, Assessed by RECIST
Description: Judged by monthly physical exam and radiographic evaluation. Patients will be considered evaluable for tumor response if they have at least two post-baseline tumor assessments at least 4 weeks apart, received study medication for 8 weeks or if they have evidence of disease progression. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 11 years
Population: All treated and eligible patients. 26 patients were not evaluable.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I/II: Oral Calcitriol, Ketoconazole, Hydrocortisone
Number analyzed (Participants) | 25
percentage of participants | 24 [9 to 45]

ADVERSE EVENTS:
Arm/Group | Phase I/II: Oral Calcitriol, Ketoconazole, Hydrocortisone
Serious Adverse Events (participants affected / at risk) | 14/51
Other Adverse Events (participants affected / at risk) | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I/II: Oral Calcitriol, Ketoconazole, Hydrocortisone (N=51)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cervical cord compression (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Visual field defect (Nervous system disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I/II: Oral Calcitriol, Ketoconazole, Hydrocortisone (N=51)
Anaemia (Blood and lymphatic system disorders) | 8 (8)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 7 (7)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Lip dry (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 28 (28)
Vomiting (Gastrointestinal disorders) | 18 (18)
Asthenia (General disorders) | 3 (3)
Chest discomfort (General disorders) | 1 (1)
Fatigue (General disorders) | 24 (24)
Gait disturbance (General disorders) | 2 (2)
Influenza like illness (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Pain (General disorders) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 3 (3)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 7 (7)
Blood alkaline phosphatase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1)
Blood calcium abnormal (Investigations) | 1 (1)
Blood calcium increased (Investigations) | 1 (1)
Blood creatine increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 23 (23)
Blood phosphorus (Investigations) | 1 (1)
Blood phosphorus increased (Investigations) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Blood potassium increased (Investigations) | 1 (1)
Carbon dioxide abnormal (Investigations) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 1 (1)
Glycosylated haemoglobin increased (Investigations) | 1 (1)
Haematocrit decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 2 (2)
International normalised ratio increased (Investigations) | 1 (1)
Low density lipoprotein increased (Investigations) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1)
Weight decreased (Investigations) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 28 (28)
Hyperglycaemia (Metabolism and nutrition disorders) | 8 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 4 (4)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1)
Cranial nerve disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Somnolence neonatal (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 3 (3)
Dysuria (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 3 (3)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Cataract operation (Surgical and medical procedures) | 1 (1)
Hot flush (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes